CLINICAL TRIAL: NCT05455619
Title: Study to Assess the Safety and Efficacy of Evexomostat (SDX-7320) in Combination With A PI3K or Akt Inhibitor Plus Fulvestrant in Patients With HR+, HER2-, Metastatic Breast Cancer With PI3K Pathway Alteration(s)
Brief Title: Evexomostat Plus PI3K or AKT Inhibitor and Fulvestrant in Patients With a PI3K Alteration and HR+/Her2- Breast Cancer
Acronym: Amelia-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SynDevRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDX-0103
Record Dates: First submitted 2022-06-22; First posted 2022-07-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: HR+/HER2-negative Breast Cancer; Metastatic Breast Cancer
Keywords: hyperglycemia; insulin; glucose; SDX-7320; fulvestrant; apelisib; PIK3CA mutation; evexomostat; HR+ Her2- metastatic breast cancer; hyperinsulinemia; capivasertib; AKT; PTEN
MeSH Terms: conditions — Breast Neoplasms; Hyperglycemia; Insulin Resistance; Hyperinsulinism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Evexomostat (Experimental): Each subject will receive repeat doses (C1, C2…) for 28-day cycles. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: Evexomostat

INTERVENTIONS:
Drug: Evexomostat — Evexomostat (SDX-7320) is a synthetic copolymer-drug conjugate of a novel MetAP2 inhibitor.
  Other Names: SDX-7320

SUMMARY:
This is a Phase 1b/2, open-label, parallel-arms pilot study in men and post-menopausal women with hormone receptor positive (HR+), HER2- advanced or metastatic breast cancer with an alteration in the PI3K pathway, including a mutation of the PIK3CA gene, PTEN loss, or AKT1 mutation, designed to determine the safety of evexomostat (SDX-7320) plus standard of care treatment alpelisib (BYL-719) or capivasertib and fulvestrant (each combined, the 'triplet therapy'), to measure the severity and number of hyperglycemic events, and to assess clinical, anti-tumor benefit of the triplet therapy.

The purpose of this study is:

* to characterize the safety of the triplet drug combination consisting of either alpelisib or capivasertib (per the treating oncologist's choice) and fulvestrant plus evexomostat,
* to test whether evexomostat, when given in combination with either alpelisib or capivasertib and fulvestrant will reduce the number and severity of hyperglycemic events and/or reduce the number or dose of anti-diabetic medications needed to control the hyperglycemia for metabolically normal patients and those deemed at risk for capivasertib and alpelisib-induced hyperglycemia (insulin resistance, as measured by HOMA-IR, baseline elevated HbA1c or well-controlled type 2 diabetes), and
* to assess preliminary anti-tumor efficacy for each combination and changes in key biomarkers and quality of life in this patient population.

DETAILED DESCRIPTION:
Phosphoinositide 3-kinase (PI3K) pathway alterations frequently occur in breast cancer, conferring growth advantages to cancer cells via increased catalytic activity of various related proteins, such as protein kinase B (AKT) or via the loss of function of the negative regulator phosphatase and tensin homolog (PTEN) (He 2021). Of these alterations, the PIK3CA gene is most frequently mutated, leading to disease aggressiveness and patient mortality. Currently approved treatments targeting this pathway include alpelisib, a small molecule that inhibits the activity of the PIK3CA gene product PI3Kα, and capivasertib, a small molecule that targets the AKT protein. Both molecules have demonstrated similar clinical benefit in cancer patients with genetic alterations that activate the PI3K/Akt/ mammalian target of rapamycin (mTOR) pathway (André 2019, Turner 2023). However, hyperglycemia, a toxicity associated with PI3K and/or Akt inhibition, leads to hyperinsulinemia, re-activating the pathway and thereby limiting each drug's clinical efficacy. Management of hyperglycemia is important to ensure patients receive optimal anti-tumor therapy (Rugo 2020). Restoring insulin sensitivity and reducing levels of insulin have been suggested as ways to blunt the hyperglycemia associated with drugs that inhibit this pathway and have been reported to improve their efficacy (Hopkins 2018, Crouthamel 2009).

The purpose of this study is

* to characterize the safety of the triplet drug combination consisting of either alpelisib or capivasertib (per the treating oncologist's choice) and fulvestrant plus evexomostat,
* to test whether evexomostat, when given in combination with either alpelisib or capivasertib and fulvestrant will reduce the number and severity of hyperglycemic events and/or reduce the number or dose of anti-diabetic medications needed to control the hyperglycemia for metabolically normal patients and those deemed at risk for capivasertib and alpelisib-induced hyperglycemia (insulin resistance, as measured by HOMA-IR, baseline elevated HbA1c or well-controlled type 2 diabetes), and
* to assess preliminary anti-tumor efficacy for each combination and changes in key biomarkers and quality of life in this patient population.

This is a Phase 1b/2, open-label, parallel-arms pilot study in men and post-menopausal women with hormone receptor positive (HR+), HER2- advanced or metastatic breast cancer with an alteration in the PI3K pathway, including a mutation of the PIK3CA gene, PTEN loss, or AKT1 mutation, designed to determine the safety of evexomostat (SDX-7320) plus standard of care treatment alpelisib (BYL-719) or capivasertib and fulvestrant (each combined, the 'triplet therapy'), to measure the severity and number of hyperglycemic events, and to assess clinical, anti-tumor benefit of the triplet therapy.

The study will consist of a 14-day pre-treatment phase of evexomostat plus fulvestrant starting on C1D1 before adding either alpelisib or capivasertib on C1D15. The Triple Therapy treatment schedule is summarized in the following table. Tumor assessments will be conducted as a function of when the triplet therapy starts.

Up to 52 patients for each combination arm may be enrolled, starting with dose-escalation cohorts of up to 6 patients for each combination arm. Once the maximum tolerated dose (MTD) of the triplet therapy has been defined for each combination, additional patients will be enrolled until a total of up to 20 patients have completed at least two cycles of the triplet therapy at that dose and combination. If warranted, up to an additional 20 patients may be enrolled to further characterize the safety profile and/or anti-tumor effect of each triplet therapy.

The planned escalation scheme starts at an evexomostat dose of 36 mg/m2 (one dose below the monotherapy MTD of 49 mg/m2) in combination with either alpelisib or capivasertib and fulvestrant given at the marketed doses. Based on aggregate safety data from the first two cycles of the first 6 patients across each triplet combination, and in the absence of ≥ 2 dose-limiting toxicities (DLTs as defined herein), the Safety Review Committee (SRC), in consultation with the Sponsor and the Investigator(s), may increase the evexomostat dose for the next cohort to 49 mg/m2. In the presence of ≥2 DLTs, the SRC may decrease the evexomostat dose to 27 mg/m2 and may adjust the dose of either alpelisib or capivasertib if warranted. The dose of fulvestrant will not be adjusted. If the evexomostat dose of 49 mg/m2 is determined by the SRC not to be tolerable in combination with either alpelisib or capivasertib and fulvestrant, then current and future patients for only their respective combination treatment will receive evexomostat at 36 mg/m2.

Patients will remain on study for up to 7 cycles to characterize the safety and tolerability of the triplet therapy as well as to capture initial efficacy data (e.g., progression-free survival [PFS] following 6 months of the triplet therapy). Patients will be allowed to continue on the triplet therapy if they are receiving clinical benefit, including stable disease, as determined by their treating oncologist.

ELIGIBILITY:
Inclusion:

1. Patient is an adult male or postmenopausal female ≥18 years old at the time of informed consent(s) and has signed informed consent(s) before any trial related activities and according to local guidelines.
2. Patient with histologically and/or cytologically confirmed diagnosis of HR+, HER2- breast cancer, as determined by the local laboratory.
3. Patient has identified PI3K pathway alteration, defined as a PIK3CA mutation or PTEN loss or an AKT1 mutation using a Food and Drug Administration (FDA)-approved test, as determined either during Screening or was previously determined to have the alteration as evidenced by written documentation.
4. Patient has locally advanced (not amenable to curative therapy or metastatic) breast cancer meeting any of the following categories:

   * Relapsed disease, not amenable to curative therapy, with documented evidence of progressive disease (PD) following receipt of both (neo) adjuvant endocrine therapy and a CDK 4/6 inhibitor therapy (either alone or in combination with endocrine therapy) in the early stage or metastatic setting.
   * Newly diagnosed advanced breast cancer, with relapsed disease (i.e., documented evidence of PD) while receiving or after endocrine therapy plus a CDK 4/6 inhibitor.
5. Patient has measurable disease per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

   For bone lesions, lytic bone lesions or mixed lytic-blastic lesions, with identifiable soft tissue components, that can be evaluated by cross-sectional imaging techniques such as computed tomography (CT) or magnetic resonance imaging (MRI) can be considered as measurable lesions if the soft tissue component meets the definition of measurability per RECIST 1.1. Blastic bone lesions are non-measurable.

   For bone metastases only (without measurable lesions), patients may be accrued to the safety Cohorts only.
6. Patient has an Eastern Cooperative Oncology Group Performance Status (ECOG-PS) ≤1
7. Patient has a Screening fasting plasma glucose (FPG) level ≤140 mg/dL (7.7 mmol/L) and an HbA1c ≤6.4% (47 mmol/mol) for those taking alpelisib, or an HbA1c <8% (64 mmol/mol) for those taking capivasertib.
8. Patient has a body mass index (BMI) ≥ 20 kg/m2.
9. Patient is male or postmenopausal female. Postmenopausal is defined as any of the following:

   * ≥45 years of age and has not had menses for >2 years.
   * Amenorrheic for >2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation.
   * Post hysterectomy with oophorectomy. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. In case of oophorectomy alone, hormone level assessment (follicle-stimulating hormone, estradiol) will be done locally at Screening to confirm postmenopausal status. Patients who are on ovarian function suppression also qualify.
10. Patient is allowed prior fulvestrant treatment, provided they remain eligible for fulvestrant treatment. Patients whose disease progressed while receiving fulvestrant monotherapy are not allowed.
11. Patient is allowed prior mTOR or PI3K inhibitor treatment for patients otherwise eligible for capivasertib treatment. Likewise, patient is allowed prior mTOR or AKT treatment if they are otherwise eligible for alpelisib treatment.
12. Patient is allowed up to one (1) prior chemotherapy for their metastatic disease.
13. Patient agrees to, and is willing and able to arrive at the hospital/clinic in a fasted state (>8 hours) on designated fasting days.
14. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

    * Platelet count ≥140×109/L
    * In absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×the upper limit of normal (ULN). If the patient has liver metastases, ALT and AST ≤5×ULN.
    * Total bilirubin ≤1.5×ULN except for patient with Gilbert's syndrome who may only be included if the total bilirubin is ≤3.0×ULN or direct bilirubin ≤1.5×ULN.
    * Fasting serum amylase ≤2×ULN.
    * Fasting serum lipase ≤1.5×ULN.
    * Hemoglobin ≥ 9 g/dL.
    * Absolute neutrophil count (ANC) ≥1500/mL.
    * Creatinine clearance ≥ 50 mL/min using either the Cockcroft-Gault equation or the CKD-EPI formula for calculation of eGFR, or has chronic kidney disease (CKD) grade ≤1 as evidenced by a treating nephrologist. Alternatively, a 24-hour urine test can be performed to confirm renal sufficiency.
    * Albumin ≥ 3.5 gm/dL.
15. Patient is able to take oral medications.

Exclusion:

1. Patient has inflammatory breast cancer at screening.
2. Patient has known primary brain malignancy, active brain metastasis or active central nervous system pathology or is considered by the Investigator to be neurologically unstable. Furthermore, patients must not have received corticosteroids within 4 weeks of study entry and must have unchanged brain CT or MRI findings for at least two months prior to screening.
3. Patient has a known hypersensitivity to evexomostat, fulvestrant, alpelisib, or capivasertib, or to any of their excipients.
4. Patient has an established diagnosis of type 1 diabetes mellitus or uncontrolled (based on fasting plasma glucose [FPG] >140mg/dL or HbA1c ≥6.5% for patients assigned alpelisib) or HbA1c for patients assigned to capivasertib, type 2 diabetes or has taken insulin in the 4 weeks prior to C1D1.
5. Patient has had major surgery within 30 days or minor surgery within 14 days prior to the first study drug dose, or has not recovered from major side effects from prior surgery.
6. Patient has ongoing toxicities related to prior anti-cancer therapies that have not resolved to Grade 0 for bone marrow toxicities or ≤Grade 1 for other toxicities, per National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v.5.0), with the exception of alopecia.
7. Patient has a Child Pugh score of B or C.
8. Patient has uncontrolled human immunodeficiency virus (HIV) infection.
9. Patient has received radio therapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to enrollment, and who has not recovered to ≤Grade 1 from related side effects of such therapy (with the exception of alopecia) and/or from whom ≥25 percentage of bone marrow was irradiated.
10. Patient has a concurrent malignancy other than breast cancer or had a malignancy other than breast cancer within 2 years of enrollment, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
11. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the drug alpelisib or capivasertib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, gastric bypass or small bowel resection) based on Investigator discretion.
12. Patient has currently documented or unresolved pneumonitis/interstitial lung disease (the chest computed tomography [CT] scan performed before start of study treatment for the purpose of tumor assessment should be reviewed to confirm that there are no relevant pulmonary complications present).
13. Patient is currently receiving any of the following medications and cannot be discontinued at least 7 days prior to the start of the treatment:

    * Strong cytochrome P450 3A4 (CYP3A4) inducers
    * Inhibitors of breast cancer resistance protein (BCRP)
    * Sulfonylurea-based anti-diabetic drugs (e.g., glipizide, glyburide, etc.)
14. Patient has a history of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis.
15. Patient has unresolved osteonecrosis of the jaw (unless they are being considered for treated with capivasertib - i.e., this exclusion is only for patients being considered for alpelisib).
16. Patient has a history of severe cutaneous reaction, such as Stevens-Johnson Syndrome (SJS), erythema multiforme (EM), toxic epidermal necrolysis (TEN), or drug reaction with eosinophilia and systemic symptoms (DRESS).
17. Patient is currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment. Note: The following uses of corticosteroids are permitted: single doses (PO or IV), topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
18. Patient is nursing (lactating) or pregnant confirmed by a positive serum (hCG) test prior to initiating study treatment.
19. Patient participated in a prior investigational study within 21 days prior to the start of study treatment or within 5 half-lives of the investigational product, whichever is longer.
20. Patient has any other concurrent, severe and/or uncontrolled medical condition that would, in the Investigator's judgement, contra-indicate patient participation in the clinical study (e.g., chronic active hepatitis, severe hepatic impairment, recent cardiac events, uncontrolled heart disease)
21. Patient is not able to understand nor to comply with study instructions and requirements, including fasting requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 48 months
  Safety and tolerability profile will be assessed by Common Terminology Criteria for Adverse Events v5.0 and summarized by type, frequency, and severity of adverse events of evexomostat dosed in combination with alpelisib plus fulvestrant
Hyperglycemic Events | Up to 42 months
  Severity, number, and proportion of patients with hyperglycemic events

SECONDARY OUTCOMES:
Anti-tumor activity | 6 months
  Number of patients without disease progression
Glucose control | Up to 42 months
  Number and type of anti-diabetic agents needed for glucose control will be measured
Leptin activity | Up to 42 months
  Changes from baseline in plasma levels of fasting leptin will be measured
Adiponectin activity | Up to 42 months
  Changes from baseline in plasma levels of fasting adiponectin will be measured
Angiogenic activity (bFGF/FGF2) | Up to 42 months
  Changes from baseline in plasma levels of angiogenic biomarkers (bFGF/FGF2, VEGFC) will be measured
Angiogenic activity (VEGFC) | Up to 42 months
  Changes from baseline in plasma levels of angiogenic and tumor biomarkers will be measured
Insulin resistance | Up to 42 months
  Changes from baseline in patients at risk for hyperglycemia using the homeostatic model assessment for insulin resistance (HOMA-IR) score of insulin resistance. HOMA-IR score is calculated as follows: (fasting serum insulin (μU/ml) × fasting plasma glucose (mmol per liter)/22.5).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Team, Study Director — SynDevRx, Inc.
Locations (10):
- United States (10):
  - Loma Linda University Cancer Center, Loma Linda, California
  - Hoag Memorial Hospital Presbyterian, Newport, California
  - SHARP Healthcare, San Diego, California
  - Miami Cancer Institute at Baptist Health, Miami, Florida
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Trinity Health, Ypsilanti, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Doctors Hospital of Laredo, Laredo, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rugo HS, Andre F, Yamashita T, Cerda H, Toledano I, Stemmer SM, Jurado JC, Juric D, Mayer I, Ciruelos EM, Iwata H, Conte P, Campone M, Wilke C, Mills D, Lteif A, Miller M, Gaudenzi F, Loibl S. Time course and management of key adverse events during the randomized phase III SOLAR-1 study of PI3K inhibitor alpelisib plus fulvestrant in patients with HR-positive advanced breast cancer. Ann Oncol. 2020 Aug;31(8):1001-1010. doi: 10.1016/j.annonc.2020.05.001. Epub 2020 May 13. PMID 32416251
- [Result] Rugo HS, Lacouture ME, Goncalves MD, Masharani U, Aapro MS, O'Shaughnessy JA. A multidisciplinary approach to optimizing care of patients treated with alpelisib. Breast. 2022 Feb;61:156-167. doi: 10.1016/j.breast.2021.12.016. Epub 2021 Dec 27. PMID 35016012